CLINICAL TRIAL: NCT07387679
Title: Comparison of Myo-inositol Versus Metformin for Treating Obesity in Patients With Polycystic Ovarian Syndrome
Brief Title: Myo-inositol Versus Metformin in Patients With Polycystic Ovarian Syndrome to Treat Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muhammad Aamir Latif (Other)
Responsible Party: Sponsor-Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Organization: RESnTEC, Institute of Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dr-Ayesha-BVH
Record Dates: First submitted 2026-01-26; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Polycystic Ovarian Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Inositol; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group-A (Experimental): Women were given tablet myo-inositol 1 gm twice a day for 3 months.
  Interventions: Drug: Myo-inositol
- Group-B (Experimental): Women received metformin 250 mg three times daily for 3 months.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Myo-inositol — Women were given tablet myo-inositol 1 gm twice a day for 3 months.
  Arms: Group-A
Drug: Metformin — Women received metformin 250 mg three times daily for 3 months.
  Arms: Group-B

SUMMARY:
There are considerable gaps in the comparative effectiveness and tolerability of myo-inositol and metformin for treating obesity in patients with polycystic ovarian syndrome (PCOS). The current study aimed to give insights comparing myo-inositol versus metformin for treating obesity in patients with PCOS.

DETAILED DESCRIPTION:
A review of the literature reveals inconsistent outcomes of myo-inositol vs metformin in the treatment of obesity and metabolic disorders in patients with PCOS, with comparable results and myo-inositol frequently demonstrating superior tolerability and reduced gastrointestinal side effects relative to metformin. When treating obesity in women with PCOS, practicing gynecologists would be able to select more appropriate medications by gathering data from local contexts. It will lessen psychological consequences associated with obesity, such as discrimination, stigma, low self-esteem, and poor quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18-45 years
* Diagnosed case of PCOS for more than 6 months of duration

Exclusion Criteria:

* Women with hyperprolactinemia or hypothyroidism (on history & medical record review)
* Adrenal hyperplasia or Cushing's syndrome (on history & medical record review)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-11-29 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Reduction in body mass index | 3 months
  A reduction in the body mass index with respect to baseline was taken as efficacy of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Gul, Principal Investigator — Bahawal Victoria Hospital/Quid-e-Azam Medical College, Bahawalpur; Shehnaz Anwar, FCPS, Study Director — Bahawal Victoria Hospital/Quid-e-Azam Medical College, Bahawalpur
Locations (1):
- Bahwal Victoria Hospital, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Data can be shared on a reasonable request.